CLINICAL TRIAL: NCT06642220
Title: Ablative Yttrium-90 Radioembolization Therapy for Non-Metastatic Renal Cell Carcinoma (ARRCC Trial)
Brief Title: Ablative Radioembolization of Renal Cell Carcinoma Trial
Acronym: ARRCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Derek W. Cool (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Derek W. Cool, Principal Investigator, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRCC 2025-1
Record Dates: First submitted 2024-10-06; First posted 2024-10-15 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Carcinoma (RCC); Radioembolization
Keywords: renal cell carcinoma; radioembolization; selective internal radiation therapy (SIRT); Y-90; Transarterial radioembolization (TARE); RCC
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Y-90 radioembolization treatment arm (Experimental): Patients with non-metastatic renal cell carcinoma (RCC) that is > 4 cm without local invasion (i.e. T1b or T2) who are poor candidates for surgery will have their tumors treated with transarterial radioembolization with Y-90 glass spheres.
  Interventions: Device: Y-90 Selective Internal Radiation Therapy (SIRT)

INTERVENTIONS:
Device: Y-90 Selective Internal Radiation Therapy (SIRT) — Y-90 radioembolization will be performed using glass spheres to treat non-metastatic RCC within the kidney.

SUMMARY:
Renal cell carcinoma (RCC), the most common type of kidney cancer, is typically treated with surgery; however, there is no established therapy for patients who are not surgical candidates and who have tumours greater than 4.0 cm in size. Selective internal radiation therapy (SIRT) or radioembolization using radioactive spheres containing 90-Yttrium (Y-90) is successful at treating large tumours with high doses of radiation within the liver and might be similarly effective for treating larger RCC tumours in patients, particularly those who are not surgical candidates.

This prospective study will enroll 16 participants with RCC who are not candidates for surgery and treat them with Y-90 radioembolization using a high-dose therapy to see if it is an effective cancer therapy. Primary outcome will be RCC treatment response 1 year after the Y-90 radioembolization. Additionally, the safety, tolerability, and impact on kidney function of the therapy will be monitored for all participants. Patients will be followed for a total of 5 years to evaluate long-term outcome in cancer control and safety of the treatment.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is the 8th most common cancer in the United States with 81,610 new cases diagnosed each year. 70% of new RCC cases are localized, non-metastatic at initial diagnosis; however, the risk of disease recurrence or progression to metastatic disease is higher for larger tumors and those with higher grade disease. The standard therapy for localized renal cell carcinoma (RCC) is surgery - either partial or radical nephrectomy. However, a substantial proportion of patients with RCC are not good surgical candidates, as the average age at diagnosis is 64-year-old, and obesity, smoking, hypertension and renal disease known risk factors. Currently there are no established standard-of-care therapies for patients who are not eligible for surgery.

Unmet Clinical Need:

There is a need to establish a definitive, minimally-invasive therapy patients for with large, non-metastatic RCC who are not surgical candidates. For non-surgical candidates with small RCC (< 4 cm or T1a) percutaneous ablation has been established as an effective minimally-invasive curative therapy. However, there is currently no minimally-invasive standard of care therapy for patients with larger localized RCC (> 4 cm) who are not surgical candidates, despite these patients being at higher risk for developing metastatic disease. Percutaneous ablation can be performed in patients with tumors > 4 cm; however, long term outcomes have not been established and those ablations carry higher risks of major bleeding complications than ablation of tumours < 4 cm. SBRT has shown some promising progression-free survival data for localized RCC; however, the radiation resistance of RCC cells require higher treatment doses to achieve cytotoxic effect. The achievable therapeutic dose of SBRT is currently limited to 30-60 Gy, often due to required reductions in the externally delivered dose to protect the commonly adjacent radiosensitive colon and/or small bowel that routinely abut the kidney.

Selective internal radiation therapy (SIRT) or Yittrium-90 (Y-90) radioembolization is an endovascular therapy whereby beads loaded with the radioactive Yittrium-90 atom are injected through a catheter into the artery or arteries supplying the tumor to deliver the radiation dose internally. Radioactive decay of the Y-90 atom within the tumor's arterial bed, deposits radiation dose within 2.5 mm (maximum 11 mm) of the bead location. As such, the internal delivery of radiation, rather than external delivery of SBRT, allows for higher doses to be delivered to the tumour without exposing adjacent vulnerable organs to significant dose. Y-90 radioembolization has great success treating hepatocellular carcinoma (HCC) in the liver, commonly achieving tumor dose levels that are nearly ten times higher than SBRT (e.g. 300-500 Gy vs. 40-50 Gy). Furthermore, it has become a standard of care therapy for HCC with recent inclusion in the major international treatment guidelines. Y-90 tumor dosage of >400 Gy is the typical target with one major explant study showing complete pathological necrosis of HCC tumors when this dose was achieved8.

RCC is a good potential disease target for Y-90 radioembolization as RCC is commonly hypervascular (similar to HCC) and the kidney is an end organ typically supplied by a single renal artery. Furthermore, the radioresistant tumour biology requires high radiation doses to achieve oncologic effect, which may be best achieved with the internal radiation delivery approach.

Existing Safety Data of Y-90 in the kidney:

Health Canada approval of Y-90 radioembolization is currently only for treatment of malignancies in the liver, where it is currently a standard of care therapy for treatment of HCC. The safety of Y-90 radioembolization in the kidney has been shown in preclinical studies as well as the RESIRT Phase I trial, which is the first and only human clinical trial of Y-90 radioembolization for RCC. The 21-patient RESIRT dose-escalation study had a heterogeneous patient population with both metastatic and non-metastatic RCC. The safety study showed no dose-limiting toxicity or reduction in renal function for treatment between 75-300 Gy; however, the secondary outcome of treatment response showed partial response in only 10% of patients without any complete response. The limited treatment response is potentially related to the administered dose being lower than the 400 Gy target used in the liver for complete pathologic necrosis. For HCC, complete pathologic necrosis from Y-90 SIRT requires an achieved tumour dose of ≥400 Gy. Within the liver, Y-90 administration of tumour doses ranging between 500-1000 Gy have been tolerated without serious adverse events.

Given the known radioresistance of RCC, it is reasonable to expect that a similar or higher dose than HCC would be required to achieve an ablative therapy (i.e. ≥ 400 Gy). The RESIRT trial used resin beads for Y-90 delivery (SIRspheres, Australia) and arterial bed stasis (not permitting additional bead administration) occurred in 52% of the treated patients, which might have limited higher achievable RCC doses. Glass-sphere beads loaded with Y-90 (Therasphere, Boston Scientific) will be used instead of resin, which have higher Y-90 radiation activity per bead than the resin counterparts (2,500 Bq/bead vs. 50 Bq/bead). The higher activity per bead should overcome the maximum dose limitation in the RESIRT trial to achieve the 400+ Gy dose likely required to for complete pathologic necrosis. This is supported by a recent case report where radioembolization with Y-90 loaded on glass spheres achieved complete tumor response after delivering 1,050 Gy into a 1.5 cm RCC without any reported adverse events.

Planned Study:

A single-centre, phase II clinical trial is proposed to evaluate the oncologic efficacy of Y-90 radioembolization treatment within the kidney for patients with large (>4.0 cm), non-metastatic (localized) RCC who are not candidates or refuse the standard of care surgery. It is proposed that Y-90 radioembolization therapy with an ablative dose (400-600 Gy) into RCC within the kidney will achieve positive oncologic response and be tolerated clinically.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate and provide written consent
* Patients 18 years of age and older
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2
* Biopsy confirmed RCC > 4.0 cm and no renal vein or IVC involvement (T1b or T2 disease)
* Not suitable for or declining standard of care nephrectomy or partial nephrectomy
* Adequate hepatic function, defined by the following laboratory results:
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN) (or ≤5 × ULN if presence of liver metastases)
* Total bilirubin ≤3 × ULN
* Serum albumin ≥3.0 g/dL unless prothrombin time (PT) is within the normal range
* Adequate hematologic function, defined by the following laboratory results:
* Hemoglobin concentration ≥8.0 g/dL
* Absolute neutrophil count (ANC) ≥1000 cells/µL (≥1000 cells/mm3 )
* Platelets >50 × 109 /L (100 × 103 /mm3 )
* For women of childbearing potential (WOCBP):
* Negative serum pregnancy test within 48 hours prior to the first dose of study treatment
* Agreement to use barrier contraception and a second form of highly effective contraception (Clinical Trials Facilitation Group [CTFG] 2020) while receiving study treatment and for 7 months following their last dose of study treatment. Alternatively, total abstinence is also considered a highly effective contraception method when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Sexually active male subjects must use a condom during intercourse while receiving treatment and for at least 120 days after the last dose of the study treatment and should not father a child during this period.
* Male study subjects whose sexual partners are WOCBP must also agree to use a second form of highly effective contraception (CTFG 2020) while receiving 90Y and for at least 4 months following their last dose. Alternatively, total abstinence is also considered a highly effective contraception method when this is in line with the preferred and usual lifestyle of the subject.
* Vasectomized men are also required to use a condom during intercourse, including with a male partner, to prevent delivery of the drug via seminal fluid.

Exclusion Criteria:

* Evidence of metastatic disease on CT or MRI
* Severely impaired renal function (GFR ≤ 30 mL/min/1.73m²) and not on dialysis
* Bilateral RCC without plan for definitive therapy of the contralateral lesion
* RCC that is locally recurrent at prior surgery or ablation site (new location in same or contralateral kidney is permitted)
* Prior or concurrent kidney radiation therapy or systemic immunotherapy/TKI
* Lung shunt with estimated lung radiation dose > 30 Gy for single dose or > 50 Gy total.
* Planning angiogram cone beam CT from all accessible feeding arteries shows lack of perfusion to all or portions of the RCC tumour such that, in the investigator's opinion, Y-90 radioembolization would result in substantial RCC tumour being untreated or receive an inadequate dose.
* Contraindication to arterial renal angiogram, or both CT and MRI contrast medium
* History of severe allergy to CT contrast medium or any study product ingredients that cannot be managed medically
* History of chronic lung disease with baseline oxygen saturation < 90% or requiring home oxygen therapy.
* Congestive heart failure with ejection fraction < 40%
* Presence of active infection, defined by the investigator as clinically significant.
* Any chronic condition that is severe or unstable and, in the opinion of the investigator, would put the patient at unacceptable risk of adverse event related to the Y-90 radioembolization procedure. Such conditions include but are not limited to: unstable angina, congestive heart failure, interstitial lung disease, severe gastrointestinal disease with diarrhea.
* Life expectancy > 1 year
* Pregnant or breast-feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Oncologic tumor response at 12 months | From treatment until 12 months follow-up imaging
  Assessment the cancer treatment response within the 12 months after treatment. Oncologic response will be based on the modified RECIST (mRECIST) criteria.

SECONDARY OUTCOMES:
Treatment-related Adverse Events | Evaluated from Y-90 therapy until 30 days, 1 year & 5 year follow-up
  Clinician assessment will occur at 4-weeks, 3-months, 6-months & 12-months post-treatment and annually to 5 years. All adverse events will be categorized and graded based on Common Terminology Criteria for Adverse Events (CTCAE) grading system. All adverse events will be further classified based on relatedness to either a) the Therapeutic Intervention and b) Y-90 Radiation Dose by the following: a) unrelated, b) unlikely to be related, c) possibly related, d) probably related, e) definitely related.
  Therapeutic Intervention: Includes all procedure-related adverse events during the planning angiogram or Y-90 therapy procedures (all Y-90 Radiation Dose adverse events included as well).
  Y-90 Radiation Dose: Subset of Therapeutic Intervention that includes only those adverse events related to the Y-90 radiation therapy. Examples of dose-related events might include post-procedure fatigue/malaise, radiation colitis, acute kidney injury not related to a catheter arterial injury.
Safety and tolerability of ablative doses (400-600 Gy) of Y-90 spheres administered in the kidney | Evaluated from Y-90 therapy until 30 days, 1 year & 5 year follow-up
  Tolerability of the radiation will be characterized by dose-limiting toxicity (DLT) events. The DLT review period will be 30 days after Y-90 procedure. Any serious adverse event that is possibly, probably or definitely related to Y-90 Radiation Dose will be classified as a dose-limiting toxicity (DLT) event. Complications related only to catheter arterial embolization procedure (example puncture site bleeding, artery dissection, etc) or the planning angiogram will not be considered a DLT. Greater > 1 in 6 patients experiencing DLT events will declare the maximally administered dose and require a reduction in the target dose to 300 Gy.
  If no DLT events occur during the DLT review period for the first three patients or 1 in the first 6 patients, then the tumour target dose for future participants can be increased up to a maximum of 600 Gy (range 400-600 Gy) at the treating physician's discretion.
Impact on global renal function | Will be evaluated at the time of Y-90 therapy as well as after Y-90 therapy at 3 months (10-16 weeks), 6 months (24-30 weeks), 12 months (50-56 weeks), & 2-, 3-, 4-, 5-years time points
  Assessment of global renal function will be based on the glomerular filtration rate (GFR), calculated using the CKD-EPI Creatinine Equation (2021). GFR will be collected at baseline and at each clinical follow-up post-therapy to assess for change.
Patient-reported outcomes | Collected at enrollment and then at 7-days, 14-days, 30-days & 3 months after Y-90 therapy.
  Patient-defined symptomatic adverse events: Self-reported by participants using the National Cancer Institute's Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) form.
  Overall Side Effect Impact: Measured by the Functional Assessment of Cancer Therapy-GP5 (FACT-GP5) question from the FACT-G questionnaire - "I am bothered by side effects of treatment". Pain intensity measured by 11-point Numerical Pain Rating Score.
  Health-related quality of life measures: Quality of life and health utility will be self-reported using the EuroQol Group EQ-5D-5L form. This 5-level form evaluates 5 dimensions of (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and can generate a global preference-based score that can be used to estimate quality-adjusted life years (QALY) within the Canadian population context to facilitate cost-utility analysis.
Change in Split Renal Function | Will be calculated at the time of Y-90 therapy (baseline) as well as after Y-90 therapy at 3 months (10-16 weeks), 6 months (24-30 weeks), 12 months (50-56 weeks), & 2-, 3-, 4-, 5-years
  Estimation of the split renal function in all participants with two kidneys will be calculated based on established renal parenchymal volume equation calculated from the CT or MR scans. Changes in the split renal function following therapy will be collected at each imaging follow up
Progression free survival out to 5 years | Greater than 1 year after Y-90 therapy, up to 5 years post therapy.
  Progression-free survival will be evaluated based on the modified RECIST (mRECIST) criteria.
Metastasis-free survival out to 5 years | Greater than 1 year after Y-90 therapy, up to 5 years post therapy
  Metastasis-free survival oncologic response will be calculated.
Overall survival out to 5 years | Greater than 1 year after Y-90 therapy, up to 5 years post therapy
  Overall survival will be calculated.
Local Progression free survival out to 5 years | Greater than 1 year after Y-90 therapy, up to 5 years post therapy.
  Local progression-free survival will be evaluated looking only at the response of the treated RCC tumor based on the modified RECIST (mRECIST) criteria. This will be evaluated out to 5 years.
Oncologic Response based on PSMA PET | scans at enrollment, and 3 months and 12 months after Y-90 therapy
  Optional Exploratory outcome - Gallium Prostate specific membrane antigen (PSMA) PET-CT be performed at baseline, 3 months and 12 months to assess the impact of Y-90 therapy on the PSMA avidity of RCC tumor. Functional imaging of PSMA PET might provide an earlier assessment of RCC tumour response as compared to the conventional contrast-enhanced CT or MRI assessment.
Change in renal volume and morphology post-therapy | From enrollment until 5-years post-therapy
  Shape-based 3D volumetric assessment of the treated kidney will be evaluated at different time points to identify long-term changes to the kidney volume and contour shape that are potentially treatment related.
Procedure Time | Will be recorded immediately after the planning angiogram procedure and again after the Y-90 therapy procedure.
  The time of the interventional radiology procedure will be recorded. Including a) total room time (time between patient entering and leaving room) and b) total angiogram procedure time (from arterial puncture until final catheter removal) for both the planning angiogram and Y-90 therapy procedures will be recorded.
Procedure Costs | Will be recorded immediately after the planning angiogram procedure and again after the Y-90 therapy procedure.
  All procedure-related costs for the interventional radiology angiogram procedure (in CAD) will be recorded (e.g. Y-90 particles, disposable catheters, wires, total time in interventional radiology suite) for both the planning angiogram and the Y-90 therapy procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Time Frame: Beginning 3 months after publication and ending 48 months after article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Summerlin AL, Lockhart ME, Strang AM, Kolettis PN, Fineberg NS, Smith JK. Determination of split renal function by 3D reconstruction of CT angiograms: a comparison with gamma camera renography. AJR Am J Roentgenol. 2008 Nov;191(5):1552-8. doi: 10.2214/AJR.07.4023. PMID 18941100
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- [Background] MacKie S, de Silva S, Aslan P, Ladd L, Houang M, Cade D, Delprado W. Super selective radio embolization of the porcine kidney with 90yttrium resin microspheres: a feasibility, safety and dose ranging study. J Urol. 2011 Jan;185(1):285-90. doi: 10.1016/j.juro.2010.09.001. PMID 21075399
- [Background] de Silva S, Mackie S, Aslan P, Cade D, Delprado W. Histological Comparison of Kidney Tissue Following Radioembolization with Yttrium-90 Resin Microspheres and Embolization with Bland Microspheres. Cardiovasc Intervent Radiol. 2016 Dec;39(12):1743-1749. doi: 10.1007/s00270-016-1482-3. Epub 2016 Oct 14. PMID 27743088
- [Background] Reig M, Forner A, Rimola J, Ferrer-Fabrega J, Burrel M, Garcia-Criado A, Kelley RK, Galle PR, Mazzaferro V, Salem R, Sangro B, Singal AG, Vogel A, Fuster J, Ayuso C, Bruix J. BCLC strategy for prognosis prediction and treatment recommendation: The 2022 update. J Hepatol. 2022 Mar;76(3):681-693. doi: 10.1016/j.jhep.2021.11.018. Epub 2021 Nov 19. PMID 34801630
- [Background] Tong AK, Kao YH, Too CW, Chin KF, Ng DC, Chow PK. Yttrium-90 hepatic radioembolization: clinical review and current techniques in interventional radiology and personalized dosimetry. Br J Radiol. 2016 Jun;89(1062):20150943. doi: 10.1259/bjr.20150943. Epub 2016 Mar 24. PMID 26943239
- [Background] Gabr A, Kulik L, Mouli S, Riaz A, Ali R, Desai K, Mora RA, Ganger D, Maddur H, Flamm S, Boike J, Moore C, Thornburg B, Alasadi A, Baker T, Borja-Cacho D, Katariya N, Ladner DP, Caicedo JC, Lewandowski RJ, Salem R. Liver Transplantation Following Yttrium-90 Radioembolization: 15-Year Experience in 207-Patient Cohort. Hepatology. 2021 Mar;73(3):998-1010. doi: 10.1002/hep.31318. Epub 2020 Nov 7. PMID 32416631
- [Background] Kluetz PG, Slagle A, Papadopoulos EJ, Johnson LL, Donoghue M, Kwitkowski VE, Chen WH, Sridhara R, Farrell AT, Keegan P, Kim G, Pazdur R. Focusing on Core Patient-Reported Outcomes in Cancer Clinical Trials: Symptomatic Adverse Events, Physical Function, and Disease-Related Symptoms. Clin Cancer Res. 2016 Apr 1;22(7):1553-8. doi: 10.1158/1078-0432.CCR-15-2035. Epub 2016 Jan 12. PMID 26758559
- [Background] McGregor H, Laidlaw G, Johnson G. Ablative Radioembolization of a Synchronous Renal Cell Carcinoma and Hepatocellular Carcinoma. J Vasc Interv Radiol. 2023 Oct;34(10):1847-1849. doi: 10.1016/j.jvir.2023.06.028. Epub 2023 Jun 28. No abstract available. PMID 37391075
- [Background] Hamoui N, Gates VL, Gonzalez J, Lewandowski RJ, Salem R. Radioembolization of renal cell carcinoma using yttrium-90 microspheres. J Vasc Interv Radiol. 2013 Feb;24(2):298-300. doi: 10.1016/j.jvir.2012.10.027. Epub 2013 Jan 28. No abstract available. PMID 23369565
- [Background] de Souza PL, Aslan P, Clark W, Nour R, de Silva S. RESIRT: A Phase 1 Study of Selective Internal Radiation Therapy Using Yttrium-90 Resin Microspheres in Patients With Primary Renal Cell Carcinoma. Clin Genitourin Cancer. 2022 Oct;20(5):442-451. doi: 10.1016/j.clgc.2022.05.006. Epub 2022 May 18. PMID 35710899